CLINICAL TRIAL: NCT00350402
Title: Masked Faces in Parkinson Disease: A Randomized Double-blind Sham-treatment Controlled Clinical Trial of High Intensity Respiratory Muscle Strength Training (MST) for Treatment of Reduced Facial Expression in Parkinson Disease
Brief Title: Masked Faces in Parkinson Disease: Mechanism and Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS050633 (NIH); R01NS050633 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; masked faces; diminished facial expressivity; diminished facial expression; high intensity respiratory muscle strength training; MST
MeSH Terms: conditions — Parkinson Disease | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Intensity Muscle Strength Training (Active Comparator): This arm involved high intensity muscle strength training at 75% maximum inspiratory pressure (MIP). Training took place for 4 weeks, 5 days a week. Each daily session involved 5 sets of breathing exercises that required participants to take deep breaths (i.e., inspire) using use a breathing device. Settings on the breathing device were determined by obtaining the individual's maximal inspiratory pressure (MIP)using a specialized breathing gauge. The MIP was determined at the beginning of each week and the training device was adjusted and set at 75% MIP. Exercises took place in home setting, with weekly visit by staff. Participants kept daily exercise log.
  Interventions: Behavioral: Respiratory muscle strength training
- Sham MST (Sham Comparator): This arm (low intensity MST) was identical to the real intervention in all ways except that the training device was set at 5% maximum inspiratory pressure (MIP). Thus less muscle and breathing effort was required during this sham treatment.
  Interventions: Behavioral: Respiratory muscle strength training

INTERVENTIONS:
Behavioral: Respiratory muscle strength training — The Muscle Stength Training (MST)device is a mouthpiece that the participant uses to inspire against controlled resistance; Intervention involves use of this device for breathing exercises over 4 week period, 5 days a week, approximately 20 minutes/day.
  Other Names: Respiratory Training; Inspiratory Training; Expiratory Training

SUMMARY:
The purpose of this study is to examine the effectiveness of high intensity respiratory muscle strength training in treating blunted facial expression in people with Parkinson disease.

DETAILED DESCRIPTION:
Facial expressions are complex signals that last only a few minutes and are important for communicating intention, motivation, and emotional states. In humans, a variety of neurological and psychiatric conditions alter the tendency to use facial signals. One of the main symptoms of Parkinson disease (PD) is diminished facial expressivity or "masked facies," which refers to the expressionless appearance of individuals with the disorder.

Unfortunately, little progress has been made over the years regarding the basis of "masked faces" or strategies that might improve facial expressivity among individuals with PD. This is unfortunate because the particular symptom can have significant medical and social consequences ranging from misdiagnosis of depression to the misattribution of negative emotional states and motivation by family members and healthcare providers.

The goal of this trial is to study the effectiveness of a novel, behavioral treatment approach-high intensity respiratory muscle strength training (MST)-for blunting of facial expressions in people with PD. The MST device, a mouthpiece that the participant uses to inspire against resistance, may improve the strength and mobility of muscles around the mouth that are involved in forming facial expressions.

Study participation includes screening, baseline evaluations, 4 weeks of behavioral intervention, immediate post-treatment followup, and a 3-month follow-up. Participants will be randomly assigned to take part in high intensity respiratory MST, or a Sham MST. Participation in the study will last for approximately 5 months.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of idiopathic Parkinson disease
* Hoeh-Yahr Stage 1-3 when off medication
* Stable and optimal medical regimen for at least 3 months
* No previous surgical interventions for Parkinson's disease (i.e., deep brain stimulation, pallidotomy, stem cell implantation)
* Participants will include men and women between the ages of 45 and 80 years

Exclusion Criteria:

* Evidence of dementia based on neurocognitive testing
* Current or past history of major psychiatric disturbance (e.g., schizophrenia, bipolar disorder, substance abuse). Participants who are taking anti-depressants will not be excluded as long as they are not currently depressed (Beck Depression, SCID)
* Other neurologic disturbance (e.g., tumor, stroke, traumatic brain injury, epilepsy) or severe chronic medical illness (e.g., HIV, metastatic cancer)
* Presence of oro-facial dyskinesias
* Previous surgeries to the larynx that result in poor vocal fold closure and/or positive history of head and neck cancer
* History of smoking in the past 5 years
* Untreated hypertension
* Failing a baseline test of pulmonary function during baseline respiratory evaluation
* Known respiratory complications such as chronic obstructive pulmonary disease (POCD), asthma
* Previous surgical interventions for Parkinson's disease (i.e., deep brain stimulation, pallidotomy, stem cell implantation)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bowers, Ph.D., Principal Investigator — Professor and Area Head, Department of Clinical and Health Psychology, University of Florida; Christine Sapienza, Ph.D., Principal Investigator — Professor and Chair, Department of Communication Sciences and Disorders, University of Florida; Michael S. Okun, M.D., Principal Investigator — Assistant Professor, Co-Director Movement Disorders Program, Medical Director, National Parkinson Foundation, Department of Neurology; Hubert Fernandez, M.D., Principal Investigator — Associate Professor and Director of Clinical Trials, Movement Disorder Program, Department of Neurology, University of Florida
Locations (1):
- Cognitive Neuroscience Laboratory, L3-135, McKnight Brain Institute, University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parkinson participants were recruited from the University of Florida Center for Movement Disorders and Neurorestoration. Recruitment began in 2004 and ended in 2009.
Pre-assignment Details: Several participants were enrolled, but subsequently excluded (prior to randomization) when it was learned that they had medical conditions that had not initially been divulged or detected (i.e., seizure disorder, "booster" ECT for treatment of depression).
Groups:
- Inspiratory Muscle Strength Training (IMST): high intensity respiratory muscle strength training, 75% MIP
- Sham MST: Low intensity muscle strength training (5% MIP)
Period: Overall Study
Arm/Group | Inspiratory Muscle Strength Training (IMST) | Sham MST
Started | 21 | 21
Completed | 20 | 20
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inspiratory Muscle Strength Training (IMST) | Sham MST | Total
Number analyzed (Participants) | 21 | 21 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.3) | 68.4 (6.9) | 67.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Education [Mean (Standard Deviation); unit: years] — Education refers to total years in school, up to a maxium of 20 years
  years | 16.76 (2.57) | 15.52 (3.1) | 16.14 (2.88)
Dementia Rating Scale-2 [Mean (Standard Deviation); unit: Units on a scale] — The DRS-2 is a cognitive screening measure for ruling out dementia. Raw scores range from 0 to 144, where higher scores reflect better performance. Scores below 130 are associated with significant cognitive disturbance.
  Units on a scale | 140 (3.49) | 138 (4.44) | 139 (4.07)
Hoehn-Yahr Scale [Mean (Standard Deviation); unit: units on a scale] — This scale is used to stage the severity of Parkinson disease symptoms. The scale ranges from Stages 0 to 5. Higher scores (i.e., 5) reflect more severe stage of Parkinson disease.
  units on a scale | 2.1 (.301) | 2.29 (.463) | 2.19 (.397)

OUTCOME MEASURES:

1. Primary Outcome: Change in Facial Entropy Score From Baseline [Off Dopamine Medication]
Description: Primary outcome is change in entropy score from baseline to immediate completion of 4 week intervention. Entropy is a computer derived index of facial movement that is computed by quantifying changes in pixel intensity as the face moves over a series of video frames. Entropy values range from 0 up to 100. Higher scores reflect greater movement and expressivity (desired). In this condition ("off dopamine), entropy scores were obtained when participants were tested "off" their normal dopamine medications. Off-dopamine testing occurred after a 12-hour overnight washout period.
Time Frame: Baseline and 4 weeks (i.e., immediate after 4-week treatment)
Population: All participants who completed baseline, intervention, and post-testing. Two participants, one from each group, dropped out during first week of intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inspiratory Muscle Strength Training (IMST): 75% MIP: High intensity respiratory muscle strength training took place over 4 weeks, 5 days a week. Each exercise session involved sets of breathing exercises taking approximately 20 minutes/day. The inspiratory exercises involved a breathing device that required individuals to take "deep breaths" and breathe in (i.e., inspire). Settings on breathing device were determined by obtaining the individual's maximal inspiratory pressure (MIP) using a specialized breathing gauge. The MIP was determined each week, and the exercise breathing trainer was adjusted and set at 75% of the participant's MIP. Exercises took place in the home setting, with weekly visit by staff.
- Sham IMST: 5% MIP: The Sham IMST intervention was identical to the "real" intervention in all ways except that the MIP is set for 5% MIP. Thus, less muscle effort was required during the exercise training.
Arm/Group | Inspiratory Muscle Strength Training (IMST): 75% MIP | Sham IMST: 5% MIP
Number analyzed (Participants) | 20 | 20
units on a scale | 5.649 (6.66) | -1.605 (6.16)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training (IMST): 75% MIP vs Sham IMST: 5% MIP; Hypothesis: Parkinson patients assigned to high intensity IMST will show greater improvement in facial movement (entropy) relative to those undergoing Sham IMST; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; df = 38; t = 3.576; Mean Difference (Final Values) = 7.254, 95% CI 2-sided [3.147 to 11.362], Standard Error of Mean 2.028 — Treatment effect size: Cohen's D =1.142

2. Secondary Outcome: Change in Parkinson Disease Quality of Life-39 Scale (PDQ-39)
Description: The PDQ-39 is a widely used quality of life measure that is specific to Parkinson disease. Total raw score on the PDQ-39 ranges from 0 to 156. Higher scores reflect worse quality of life rating. Total score on PDQ-39 was used to compute pre-post treatment changes.
Time Frame: Baseline and 4 weeks (i.e., immediate post-intervention)
Population: Participants who completed baseline,intervention, and post-intervention testing. Two individuals, one from each group, dropped out of the study during the first week of intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inspiratory Muscle Strength Training (IMST): 75% MIP: Same as previously described. High intensity respiratory muscle strength training took place over 4 weeks, 5 days a week. Each exercise session involved sets of breathing exercises taking approximately 20 minutes/day. The inspiratory exercises involved a breathing device that required individuals to take "deep breaths" and breathe in (i.e., inspire). Settings on breathing device were determined by obtaining the individual's maximal inspiratory pressure (MIP) using a specialized breathing gauge. The MIP was determined each week, and the exercise breathing trainer was adjusted and set at 75% of the participant's MIP. Exercises took place in the home setting, with weekly visit by staff.
- Sham IMST: 5% MIP: Same as previously described. The Sham IMST intervention was identical to the "real" intervention in all ways except that the MIP is set for 5% MIP. Thus, less muscle effort was required during the exercise training.
Arm/Group | Inspiratory Muscle Strength Training (IMST): 75% MIP | Sham IMST: 5% MIP
Number analyzed (Participants) | 20 | 20
units on a scale | 1.850 (10.16) | -1.550 (17.57)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training (IMST): 75% MIP vs Sham IMST: 5% MIP; Hypothesis: Scores on PDQ-39 would show bigger change for the IMST group than the Sham treatment group. The sample size was not powered for the PDQ-39 (but rather for the primary outcome variable); Test type: Superiority or Other; p < 0.459, t-test, 2 sided; Mean Difference (Final Values) = -6.36, 95% CI 2-sided [-16.41 to 3.68], Standard Error of Mean 4.955

3. Other Pre Specified Outcome: Change From Baseline in Maximal Inspiratory Pressure (MIP)
Description: The dependent variable is the change in maximal inspiratory pressure (MIP) from baseline to immediate completion of 4-week intervention. MIP refers to how much air pressure force an individual creates by inhaling through the mouth as hard as possible. This was measured over 5-7 trials by placement of lips around a mouthpiece attached to a calibrated fluke digital pressure gauge. From these trials, an average maximum inspiratory pressure (MIP) was computed. This was done at baseline and post-treatment. Greater MIP changes correspond to greater treatment-related effects of exercise.
Time Frame: Baseline and 4 weeks (i.e., immediate after 4-week intervention)
Population: Included participants who underwent baseline, intervention, and post-treatment assessment. Two individuals dropped out during the first week of intervention, one from each intervention group. Additionally, there was faulty data, due to equipment failure for one individual in the sham group, thereby reducing N in this group to 19.
Measure: Mean (Standard Deviation); unit: units of pressure (cmH20)
Groups:
- Inspiratory Muscle Strength Training (IMST): 75% MIP: high intensity respiratory muscle strength training, 75% MIP
- Sham IMST: 5% MIP: Low intensity muscle strength training (5% MIP)
Arm/Group | Inspiratory Muscle Strength Training (IMST): 75% MIP | Sham IMST: 5% MIP
Number analyzed (Participants) | 20 | 19
units of pressure (cmH20) | 13.9 (12.16) | 3.47 (14.16)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training (IMST): 75% MIP vs Sham IMST: 5% MIP; Hypothesis: Changes in MIP following treatment would be greater for participants in the IMST versus the Sham treatment group. This is a validity check on for the IMST intervention; Test type: Superiority or Other; p < 0.018, t-test, 2 sided; t-value = 2.47, with 37 df; Mean Difference (Final Values) = 10.426, 95% CI 2-sided [1.874 to 18.978], Standard Error of Mean 4.221

4. Primary Outcome: Change in Facial Entropy Score From Baseline [On Dopamine Medication]
Description: Outcome is entropy change from baseline to immediate completion of 4 week intervention when participants remained on their normal dosage of dopamine medication. Entropy is quantitative index of facial movement that is computed from changes in pixel intensity as the face moves. Entropy values range from 0 up to 100. Higher scores reflect greater movement and expressivity. Greater expressivity is desired outcome.
Time Frame: Baseline and 4 weeks (i.e., immediate after 4-week intervention)
Population: Based on individuals who completed baseline and post-treatment assessment following 4 weeks of intervention. One individual from each treatment group dropped out during the first week of intervention and were not included in analyses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Inspiratory Muscle Strength Training (IMST): 75% MIP: Same as previously described. This intervention involves high intensity respiratory muscle strength training over 4 week period, 5 days a week, with training device set at 75% maximal inspiratory pressure (MIP). The MIP is determined weekly and the training device recalibrated to take into account changes.
- Sham IMST: 5% MIP: This intervention is identical in all ways to "real" treatment, except that training device requires less inspiratory effort. The training device is set at 5% MIP. )
Arm/Group | Inspiratory Muscle Strength Training (IMST): 75% MIP | Sham IMST: 5% MIP
Number analyzed (Participants) | 20 | 20
Units on a scale | 3.559 (9.995) | -1.569 (4.931)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training (IMST): 75% MIP vs Sham IMST: 5% MIP; Hypothesis: Facial entropy changes would be greater in IMST group than sham treatment group. Sample size was based on preliminary data suggesting total N of 40 would be adequate for detecting change in entropy (of approximately 50%); Test type: Superiority or Other; p < 0.047, t-test, 2 sided — No adjustment necessary; 38 df, t= 2.058 However, due to inequality of variance (Levine test), the adjusted p-value = <0.049, and adjusted df = 27.3; Mean Difference (Final Values) = 5.129, 95% CI 2-sided [.0834 to 10.17], Standard Error of Mean 2.492

ADVERSE EVENTS:
Time Frame: Data collected for 6 months
Arm/Group | Inspiratory Muscle Strength Training (IMST) | Sham MST
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No